CLINICAL TRIAL: NCT04533997
Title: Efficacy and Safety of Ambulatory Hypertonic Saline Therapy in Outpatient Heart Failure Units.
Brief Title: Hypertonic Saline Therapy in Ambulatory Heart Failure Unit.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Marta Cobo Marcos, Cardiologist, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SALT-HF TRIAL
Record Dates: First submitted 2020-08-23; First posted 2020-09-01 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure
Keywords: Hypertonic Saline Solution; Outpatient Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Intervention Model Description: Randomization 1:1 to treatment with a 1-hour infusion of IV furosemide plus HSS (2.6-3.4% NaCl depending on plasmatic sodium levels) versus a 1-hour infusion of IV furosemide at the same dose (125-250 mg, depending on basal loop diuretic dose).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Based on an automated online system, blinded to the physicians who evaluated the patient.
  Randomization was performed by a trained nurse in a separate room
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous furosemide (Active Comparator)
  Interventions: Drug: Intravenous furosemide
- Hypertonic saline solution plus intravenous furosemide (Experimental)
  Interventions: Drug: Hypertonic saline solution plus intravenous furosemide

INTERVENTIONS:
Drug: Hypertonic saline solution plus intravenous furosemide — Intravenous 60-minutes of hypertonic saline therapy plus furosemide:
  Furosemide:
  125 mg if home oral furosemide ≤160 mg, 250 mg if home oral furosemide > 160 mg
  Hypertonic saline solution:
  Na+ 125-134: 3.4%, Na+ 135-145: 2.6%
  Arms: Hypertonic saline solution plus intravenous furosemide
Drug: Intravenous furosemide — Intravenous 60-minutes infusion of furosemide:
  125 mg if home oral furosemide ≤ 160 mg, 250 mg if home oral furosemide > 160 mg
  Arms: Intravenous furosemide

SUMMARY:
The purpose of this study is to compare intravenous furosemide (125 to 250 mg), isolated or in combination with hypertonic saline solution (2.6% to 3.4%) in the outpatient heart failure patient. The hypothesis is that the combination therapy will increase the diuresis volume at 3 hours and improve congestion parameters at 7 days.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multicenter study of all consecutive patients with decompensated heart failure and signs of volume overload who do not require hospital admission but require intravenous diuretic for relief of congestion.

Patients meeting the inclusion criteria, with prior informed consent, will be randomized to treatment with furosemide with hypertonic saline versus isolated furosemide (control group).

Complete clinical evaluation, echocardiography, and blood and urinary tests will be performed before the treatment. After 3 hours, diuresis volume, weight and urinary parameters will be evaluated. Efficacy and safety visits will be performed at 7 and 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Previous heart failure diagnosis (according to current European Guidelines)
* Stable treatment in the previous 4 weeks (except diuretic).
* Home oral treatment of ≥80 mg of furosemide/day or equivalent (40 mg furosemide = 20 mg of torasemide).
* Transthoracic echocardiogram performed in the last year.
* Congestive signs.The presence of two of the following congestion criteria will be required: jugular pressure> 10 cm, lower limb edema, ascites, or pleural effusion
* Elevation of natriuretic peptides (NTproBNP> 1000 pg / mL or B-type natriuretic peptide> 250 pg / ml) performed in a previous period of no more than 24 hours.
* Need for intravenous diuretic therapy to relieve congestion according to the responsible physician.

Exclusion Criteria:

* Hospital admission criteria in the opinion of the responsible physician.
* Systolic blood pressure <90 mmHg or> 180 mmHg.
* Heart rate> 150 bpm or < 40 bpm
* Basal oxygen saturation less than 90%.
* Cardiogenic shock.
* Acute Pulmonary Edema.
* Clinically significant arrhythmia.
* Acute myocardial ischemia.
* Patients in hemodialysis or peritoneal dialysis program.
* Serum sodium <125 milliequivalent / L or> 145 milliequivalent / L.
* Serum potassium < 3.5 milliequivalent/ L.
* Hemoglobin < 9 g / dL
* Acute coronary syndrome or cardiological procedure in the previous 2 weeks.
* Severe uncorrected valve disease except tricuspid regurgitation.
* Moderate or severe dementia, active delirium or psychiatric problems.
* Patients in whom cardiac surgery or device implantation is planned in the following 30 days.
* Pregnancy or breastfeeding.
* Inability to give informed consent in the absence of a legal officer.
* Patients on tolvaptan.
* Inability to collect the urine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Diuresis volume (ml) | 3 hours after treatment
  Total diuresis volume after 3 hours of therapy administration

SECONDARY OUTCOMES:
Weight difference (kg) | 3 hours
  Difference of weight 3 hours after the start of treatment
Weight difference (kg) | 7 days
  Difference of weight 7 days after the start of treatment
Change in composite congestion score | 7 days
  Composite of orthopnoea (0-3), jugular venous distension (0-3), lower limb oedema (0-3). Higher score: worse congestion
Change in Inferior cava vein diameter (mm) | 7 days
  Change in Inferior cava vein diameter (mm) 7 days after treatment
Change in Number of fields with more than 3 B-lines in lung ultrasound | 7 days
  Change in Number of fields with more than 3 B-lines in lung ultrasound 7 days after treatment
Change in New York Heart Association and Visual Analogue Scale | 7 days
  Visual Analogue Scale from 0 (worst state of health) to 100 (best state of health)
Change in NTproBNP and Cancer Antigen 125 levels | 7 days
  Change in NTproBNP and Cancer Antigen 125 levels 7 days after treatment
Change in Hemoconcentration Parameters | 7 days
  Hematocrit, Albumin and total Proteins
Change in Urinary Sodium | 7 days
  Change in Urinary Sodium measured in a spot urinary sample
Adverse Events | 7 days
  Need of new intravenous diuretic (outpatient clinic or emergency department). Heart Failure hospitalization. Cardiovascular mortality. All-Cause mortality or hospitalization. Worsening of kidney function: defined as an increase in creatinine ≥ 0.3 mg / dl.
  Electrolyte abnormalities defined as hypokalemia (K+ less than 3.5 milliequivalent / L) or hyperkalemia (K+ greater than 5.5 milliequivalent /L)
Adverse Events | 30 days
  Need of new intravenous diuretic (outpatient clinic or emergency department). Heart Failure hospitalization. Cardiovascular mortality. All-Cause mortality or hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Cobo Marcos, MD, Principal Investigator — Hospital Universitario Puerta de Hierro. Madrid. Spain
Locations (14):
- Spain (14):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital de la Santa Creu i Santa Pau (Fundación Privada Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico Universitario San Carlos, Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Clínico Universitario Lozano de Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF